CLINICAL TRIAL: NCT06604715
Title: A Phase 1, First-in-Human, Open-Label, Dose Escalation Study of JNJ-87562761 in Relapsed/Refractory Multiple Myeloma
Brief Title: A Study of JNJ-87562761 in Participants With Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 87562761MMY1001; 87562761MMY1001 (Other: Janssen Research & Development, LLC); 2024-513439-25-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-09-18; First posted 2024-09-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JNJ-87562761 (Experimental): Participants will receive JNJ-87562761 during the Part 1 (Dose escalation) to determine the recommended phase 2 dose (RP2D) regimen(s). The dose will be escalated sequentially until the RP2D regimen(s) have been identified. In Part 2 (Dose expansion) participants will receive JNJ-87562761 at the RP2D regimen(s) determined in Part 1.
  Interventions: Drug: JNJ-87562761

INTERVENTIONS:
Drug: JNJ-87562761 — JNJ-87562761 will be administered.

SUMMARY:
The purpose of this study is to determine the recommended phase 2 dose(s) (RP2D[s]) of JNJ-87562761 in Part 1 (dose escalation), and to determine the safety and tolerability at RP2D in Part 2 (dose expansion) in participants with multiple myeloma (MM) whose disease has come back after treatment (relapsed) or hasn't responded to treatment (refractory).

ELIGIBILITY:
Inclusion Criteria:

* Relapsed, refractory multiple myeloma with measurable disease defined as: (a) Serum monoclonal paraprotein (M-protein) level greater than (>)0.5 grams per deciliter (g/dL); or (b) Urine M-protein level >200 milligrams per 24 hours (mg/24 hours); or (c) Light chain multiple myeloma: serum immunoglobulin free light chain (FLC) >10 milligrams per deciliter (mg/dL) and abnormal serum immunoglobulin kappa-lambda FLC ratio
* Must have had prior therapy including a proteasome inhibitor, immunomodulatory agent and anti-CD38 therapy
* Have an eastern cooperative oncology group (ECOG) performance status of 0 to 1
* Have an estimated glomerular filtration rate (eGFR), of > 30 millilitres (mL)/min/1.73 meter square (m^2) computed per 2021 chronic kidney disease epidemiology collaboration (CKD-EPI) creatinine equation
* While on study treatment and for 6 months after the last dose of study treatment, a participant must: (a) Not breastfeed or be pregnant; (b) Not donate gametes (that is, eggs or sperm) or freeze for future use for the purposes of assisted reproduction; (c) Wear an external condom

Exclusion Criteria:

* Active plasma cell leukemia, Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes), or immunoglobulin light chain amyloidosis
* Prior allogeneic transplant within 6 months before the start of study treatment administration or autologous transplant within 12 weeks before the start of study treatment administration
* Live, attenuated vaccine within 4 weeks before the first dose of study treatment
* Central Nervous System (CNS) involvement or clinical signs of meningeal involvement of multiple myeloma. If either is suspected, brain magnetic resonance imaging (MRI) and lumbar cytology are required
* Non-hematologic toxicity from prior anticancer therapy that has not resolved to baseline level or to less than or equal to (<=) Grade 1 (except alopecia, tissue post-RT fibrosis, or Grade < 3 peripheral neuropathy)
* Received a cumulative dose of corticosteroids equivalent to greater than or equal to (>=) 140 mg of prednisone within the 14-day period before the start of study treatment administration
* Prior antitumor therapy in the specified time frame prior to the first dose of study treatment: (Targeted therapy, epigenetic therapy, monoclonal antibody treatment, or treatment with an investigational drug or an invasive investigational medical device or conventional chemotherapy within 21 days, gene-modified adoptive cell therapy or treatment with anti-CD38 directed therapies within 3 months, proteasome inhibitor [PI] therapy or radiotherapy within 14 days, or immunomodulatory drug (IMiD) agent therapy within 7 days)
* Following medical conditions: pulmonary compromise requiring supplemental oxygen use to maintain adequate oxygenation, human immunodeficiency (HIV) infection (participants with a detectable viral load or low CD4 count), active hepatitis B or C infection, active autoimmune disease requiring systemic immunosuppressive therapy within 6 months before start of study treatment, serious uncontrolled ongoing viral or bacterial or systemic fungal infection, cardiac conditions (myocardial infarction <=6 months prior to enrollment, New York Heart Association stage III or IV congestive heart failure, et cetera [etc.])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2027-11-03 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Dose-Limiting Toxicity (DLT) | up to approximately 3 years
  DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity or hematologic toxicity.
Part 1 and 2: Number of Participants with Adverse Events (AEs) | up to approximately 3 years
  Number of participants with AEs will be reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Part 2: Number of Participants with Clinically Significant Abnormal Laboratory Values | up to approximately 3 years
  Number of participants with clinically significant abnormal laboratory values (hematology or chemistry) will be reported.

SECONDARY OUTCOMES:
Serum Concentration of JNJ-87562761 | up to approximately 3 years
  Serum samples will be analyzed to determine concentrations of JNJ-87562761.
Pharmacokinetic (PK) Parameters of JNJ-87562761 | up to approximately 3 years
  PK parameters for JNJ-87562761 will be evaluated.
Number of Participants with Presence of Anti-JNJ-87562761 Antibodies | up to approximately 3 years
  Number of participants with presence of anti-JNJ-87562761 antibodies will be reported.
Percentage of Participants with Response | up to approximately 3 years
  Overall response is defined as a best response of partial response (PR) or better as assessed according to the International Myeloma Working Group (IMWG) 2016 response criteria.
Percentage of Participants Who Achieve Very Good Partial Response (VGPR) or Better | up to approximately 3 years
  VGPR or better response is defined as the percentage of participants who achieve a best response of VGPR or better as assessed by IMWG 2016 response criteria.
Percentage of Participants Who Achieve Complete Response (CR) or Better | up to approximately 3 years
  CR or better response is defined as percentage of participants who achieve a best response of CR or better as assessed by IMWG 2016 response criteria.
Percentage of Participants Who Achieve Stringent Complete Response (sCR) | up to approximately 3 years
  sCR is defined as the percentage of participants who achieve a best response of sCR as assessed by IMWG 2016 response criteria.
Duration of Response (DOR) | up to approximately 3 years
  DOR is defined for participants who achieve a response of PR or better as the time from the first efficacy evaluation at which the participant met all criteria for a response of PR or better to the time of first documented evidence of progressive disease or death, assessed by IMWG 2016 response criteria.
Time to Response (TTR) | up to approximately 3 years
  TTR is defined for participants who achieve a response of PR or better as the time from the first dose of study drug to the time of the first efficacy evaluation at which the participant met all criteria for a response of PR or better, assessed by IMWG 2016 response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (15):
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (5):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency